CLINICAL TRIAL: NCT03030352
Title: How to Talk so Kids Will Listen & Listen so Kids Will Talk: A Randomized Controlled Trial Assessing the Impact of the French Workshop Format in the General Population
Brief Title: Promoting Children's Mental Health: The Effects of a Parenting Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Mireille Joussemet, Associate Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MOP-130576
Record Dates: First submitted 2016-12-09; First posted 2017-01-25 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Child Development
Keywords: Child Mental Health; Parenting; Autonomy Support; How-to Parenting Program; Randomized Controlled Trial; Primary Prevention; Parental Mental Health; Child Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- How-to Parenting Program (Experimental): The How-to Parenting Program consists of seven 2 ½-hour weekly sessions. It is a manual-based program in which participants have their own exercise booklet containing parenting skills and exercises. Groups are led by 2 group leaders and formed of 6 to 10 parents.
  Interventions: Behavioral: How-to Parenting Program
- Wait-list Control Group (No Intervention): Parents assigned to the wait-list control group will receive no intervention for the duration of the trial. The How-to Parenting Program will be delivered to them the following year. This delayed participation is ethically sound, as the program does not target at-risk families.

INTERVENTIONS:
Behavioral: How-to Parenting Program — The How-to Parenting Program addresses all three key dimensions of optimal parenting; autonomy support, affiliation and structure. With weekly workshops, the How-to-Parenting Program optimizes learning by (1) linking group content with parents' needs, (2) facilitating awareness with perspective taking activities, (3) offering concrete parenting skills, (4) modeling the skills and providing practice in a predictable and non-judgmental environment, (5) emphasizing the importance of implementing these skills at home for long term behavioral change, and (6) offering tools (i.e., exercise booklet, skill summary) that facilitate information retention.
  Other Names: How to talk so kids will listen & listen so kids will talk
  Arms: How-to Parenting Program

SUMMARY:
The objectives of the How-to parenting program are 1) to improve optimal parenting style, and 2) to foster children mental health (i.e. decrease in internalized and externalized problems, and well-being). The investigators expect that parents assigned to experimental groups will show improvements in parenting over time (i.e improvements in parental affiliation, parental structure and parental attitude toward autonomy), whereas parents in control groups will not show such improvements (i.e., stable or declining parenting quality). The investigators also expect children of parents in experimental groups to experience improvements in child mental health (i.e., fewer internalized and externalized psychological problems and increased well-being), whereas children whose parents are on the wait list will not show improvements over time (i.e., stable or deteriorating mental health and well-being).

DETAILED DESCRIPTION:
Raising children is a fundamental yet challenging task. While parents are highly invested in their children's development, they also have a vast influence on it. Indeed, among environmental factors, the most widely accepted predictor of children mental health is parenting quality. Research has shown that optimal parenting is composed of three key dimensions: structure, autonomy support, and affiliation (vs. permissiveness, psychological control, rejection). For parents, providing all three key "nutriments" is not necessarily natural or easy. Indeed, it can be challenging to (1) require children to adopt socially desirable behaviors (2) without thwarting their need for self-determination, (3) while preserving a positive parent-child relationship. In addition, available parenting resources (e.g., diverse parenting books) are sometimes contradictory, abstract, and rarely tap all three important parenting dimensions. Providing the general population with concrete and complete parenting education is essential in helping parents with their important yet challenging role.

The goal of the proposed research is to evaluate a parenting program (i.e., How-to program) that addresses all three key dimensions of optimal parenting. This program is congruent with basic developmental research and with knowledge from decades of motivation research devoted to autonomy support and self-determination theory. The objectives of the How-to parenting program are 1) to improve optimal parenting style, and 2) to foster children mental health (i.e. decrease child' internal and external problems, and increase child' well-being). The investigators expect that parents assigned to experimental groups will show improvements in parenting over time, whereas parents in control groups will not show such improvements (i.e., stable or declining parenting quality). The investigators also expect children of parents in experimental groups to experience improvements in mental health, whereas children whose parents are on the wait list will not show improvements over time (i.e., stable or deteriorating mental health and well-being).

The research team will recruit participants and conduct the study in four schools per year, during four years. The How-to parenting program will be offered to parents of grade school children (5 to 12 years old). Grade schools will be recruited through Montreal school boards. Only one parent per family may participate in the study. If parents have more than one child in grade school, they will be asked to identify the one who is closest to 9 years of age and then answer questionnaires about this "targeted" child. The seven-week parenting program will be offered to the experimental groups (one per school) each spring (Years 1 to 4). Each of these 4 experimental groups will be paired with a wait list control group from the same school. Parents from these control groups will be offered the program the following year (Years 2 to 5). In total, 256 parents from different families (mothers or fathers) will be recruited in participating schools (16 parents [8 in experimental group + 8 in control group] in each of 4 schools, for 4 years). This sample size was chosen to achieve adequate power, while keeping the study feasible given participation rate.

The How-to program highlights the importance of structure and teaches parents how to provide it. Parents learn how to communicate expectations, give feedback, follow through with logical consequences and use problem solving for recurrent problems. In addition, the program perfectly captures what it means to be autonomy-supportive. Moreover, this style helps children feel better about the rules and about themselves. These new skills empower parents to exert their authority with confidence and, importantly, without guilt. Parents are then more apt at providing structure effectively and consistently. With the How-to Parenting program, parents learn how to listen and respond to their children in a way that helps children feel loved and accepted for who they are.

The How-to parenting program consists of seven 2 ½-hour weekly sessions. It is a manual-based program in which participants have their own exercise booklet containing parenting skills and exercises. Groups are led by 2 group leaders and formed of 6 to 10 parents. The format of this program optimizes learning by (1) linking group content with parents' needs, (2) facilitating awareness with perspective taking activities, (3) offering concrete parenting skills, (4) modeling the skills and providing practice in a predictable and non-judgmental environment, (5) emphasizing the importance of implementing these skills at home for long term behavioral change, and (6) offering tools (i.e., exercise booklet, skill summary) that facilitate information retention.

All parents and children will complete the same questionnaires before randomization (baseline), after the seven-week program (post-test), and again at 6-month and 1-year follow ups to assess change over time. Data will also be collected from targeted children's teachers. These teacher reports will be collected at school, at each assessment point. At follow ups, teacher reports will be provided by participating children's new teachers (i.e., in October and April of the 2nd school year). All measures (except for the control variables) are included at all four assessment times to allow change measurement. The investigators will adopt an intent-to-treat approach, as this approach increases external and internal validity.

Parenting style measures were reviewed and selected to best reflect recent conceptualizations of the three key parenting dimensions and to do so with the least overlap. Affiliation (Parental Bonding Instrument), structure (Parenting Scale), and attitude toward autonomy (How-to Parenting Skill Scale; Parental Autonomy Support Scale (P-PASS)) are assessed by parents and children. Child mental health will be assessed using a multi-source approach (parent, teacher and child reports). Parents will rate their child's internalized and externalized psychological problems (Child Behavior Checklist; CBCL). Teachers are asked to evaluate children's classroom and social problems (Teacher-Child Rating Scale; TCRS). The problem subscales of the TCRS assess internalized (I-) and externalized-(E-) problems. Teachers will also complete the competencies subscales of the TCRS, which evaluate socio-emotional competencies (i.e., frustration tolerance, task orientation and social skills).

In the present data, baseline, post-test, and 6-month and 1-year follow up measures are nested within a parent, who are nested within a parenting group. To evaluate change over time, the four assessment points (baseline, post-test, 6-month follow up, and 12-month follow up) will be treated as repeated measures using a piecewise growth hierarchical linear modelling (HLM). These analyses are chosen because they model change between each subsequent time points, which allows for rates of change to differ across time. HLM models are recommended for intervention studies in order to capture rates of change both in the intervention period and in the follow up periods. The effect of the parenting program will be evidenced by significant interactions between rates of change and experimental conditions. These interactions should reveal that optimal parenting components (H1) and child mental health indicators (H2) increase over time for participants in the experimental condition, but not for participants in the control group.

By including all three dimensions of optimal, authoritative parenting, the How-to program stands in contrast to the majority of existing parenting training programs. In general, most interventions target children already showing behavioral problems or considered at risk and focus on behavior management strategies such as planned ignoring or reinforcement. Results from a recent meta-analysis provide support for the adoption of a program that encompasses all of the three essential dimensions of optimal parenting. Indeed, results showed that programs' components that were predictive of larger effects pertained to autonomy support, affiliation and structure. Though no formal evaluation of the How-to program has been made, one early study suggested that it was associated with better familial climate and parenting practices.

This proposal is a first step toward implementing and evaluating a parenting program tailored to the promotion of children's mental health. By improving parenting, it can ameliorate children's life-course trajectories, thereby reducing mental health problems and their associated costs. By offering parenting groups, this research project includes a significant knowledge transfer component that will directly impact parents enrolled in the program. Dissemination of findings will be made in schools, by giving school principals, teachers and parents an easy-to-read summary of results. If the present randomized controlled trial and following replication trials are successful, a wider dissemination/evaluation trial will be implemented, making the program widely available to parents.

ELIGIBILITY:
Inclusion Criteria:

* Parents must have a child (5-12 years old) attending a participating grade school

Exclusion Criteria:

* Inability to communicate in the language in which the study is conducted (i.e., French)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2014-02; Primary Completion 2017-04-28 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change in parenting style assessed by parents | 1 week post-intervention, 6 months and 1 year follow-up
  Parenting Style will be assessed by a self-administered questionnaire with 3 subscales.
  Parental Bonding Scale, Parenting Structure Scale, and Parental Autonomy Support scale.
Change in children's mental health problems at home | 1 week post-intervention, 6 months and 1 year follow-up
  Parents will rate their child's I- and E- psychological problems with a questionnaire composed with the Child Behavior Checklist CBCL.
Change in children's mental health problems at school | 1 week post-intervention, 6 months and 1 year follow-up
  Teachers are asked to evaluate children's classroom and social problems with the Teacher-Child Rating Scale; TCRS. The problem subscales of the TCRS assess I- (shy-anxious) and E- (acting-out) problems.
Change in children's competencies at school | 1 week post-intervention, 6 months and 1 year follow-up
  Teachers will complete the competencies subscales of the TCRS, which evaluate children' socio-emotional competencies (i.e., frustration tolerance, task orientation and social skills).
Change in children's well-being | 1 week post-intervention, 6 months and 1 year follow-up
  Children will assess their own well-being with a self-administered questionnaire with 3 positive indicators; self-esteem, life satisfaction and positive affect.

SECONDARY OUTCOMES:
Change in parenting style assessed by children | 1 week post-intervention, 6 months and 1 year follow-up
  Children will assess change in parenting style by answering a child report questionnaire.
Change in parent's mental health problems | 1 week post-intervention, 6 months and 1 year follow-up
  Parents will assess their own mental health by rating their psychological symptoms (i.e., negative affect, PANAS; anxious and depressive symptoms, General Health Questionnaire).
Change in parent's well-being | 1 week post-intervention, 6 months and 1 year follow-up
  Parents will assess their own well-being with a self-administered questionnaire with 3 positive indicators; self-esteem, life satisfaction and positive affect.
Change in perceived parental competencies | 1 week post-intervention, 6 months and 1 year follow-up
  Parents will assess their perceived parental competencies by rating the Basic Need Satisfaction in Relationships Scale.
Change in parental guilt | 1 week post-intervention, 6 months and 1 year follow-up
  Parents will assess their guilt by rating the expanded PANAS.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Joussemet, Ph.D., Principal Investigator — Université de Montréal; Geneviève Mageau, Ph.D., Principal Investigator — Université de Montréal
Locations (1):
- University of Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Joussemet M, Mageau GA, Larose MP, Briand M, Vitaro F. How to talk so kids will listen & listen so kids will talk: a randomized controlled trial evaluating the efficacy of the how-to parenting program on children's mental health compared to a wait-list control group. BMC Pediatr. 2018 Aug 2;18(1):257. doi: 10.1186/s12887-018-1227-3. PMID 30071843
- Available data/document: Pilot Study of the How-to trial — http://link.springer.com/article/10.1007/s10826-013-9751-0